CLINICAL TRIAL: NCT00469170
Title: A Safety and Acceptability Study of a Vaginal Ring Microbicide Delivery Method for the Prevention of HIV Infection in Women
Brief Title: A Safety and Acceptability Study of a Vaginal Ring Microbicide Delivery Method
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Annalene Nel, International Partnership for Microbicides
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IPM 011
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: HIV-1; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): vaginal ring first 12 weeks & observational safety last 12 weeks
  Interventions: Device: intravaginal ring
- B (Experimental): observational safety first 12 weeks & vaginal ring last 12 weeks
  Interventions: Device: intravaginal ring

INTERVENTIONS:
Device: intravaginal ring — silicone elastomer intravaginal ring containing no drug product

SUMMARY:
The proposed study is a multi-centre, open-label crossover study to assess the safety and acceptability of a silicone elastomer vaginal ring (containing no drug) when inserted for a 12 week period in 200 healthy, sexually active women.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-35 years
* Willing and able to provide written informed consent
* HIV-uninfected and otherwise healthy
* Self-reported sexually active
* On a stable hormonal contraceptive regimen
* Regular menstrual cycle
* Willing to refrain from use of vaginal products or objects during the study

Exclusion Criteria:

* Currently pregnant or last pregnancy within 3 months prior to enrollment
* Currently breast-feeding
* Participated in any other research study within 30 days prior to enrollment;
* Symptomatic untreated vaginal infections within 2 weeks prior to enrollment
* Presence of abnormal physical finding on the vulva, vaginal walls or cervix
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction;
* Pap smear result at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation
* Unexplained, undiagnosed abnormal bleeding per vagina, bleeding per vagina during or following vaginal intercourse, or gynecologic surgery within 90 days prior to enrollment
* Any serious acute, chronic or progressive disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary measure of acceptability will be defined as the proportion of women indicating that they would use the study product if it is found to prevent HIV. | 3 months
The primary measure of safety will be the proportion of women who have abnormal observations during the pelvic/speculum examinations and the proportion of women who experience adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Annalene Nel, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (4):
- South Africa (3):
  - Reproductive Health & HIV Research Unit - Sheshisani IPM Clinic, Yeoville, Johannesburg
  - South African Medical Research Council, Durban, KwaZulu-Natal
  - Desmond Tutu HIV Foundation, Masiphumelele, Cape Town
- Kilimanjaro Reproductive Health Program, Moshi, Tanzania